CLINICAL TRIAL: NCT05327283
Title: Insight Into the Genomics of Idiopathic Premature Ovarian Insufficiency
Brief Title: Investigation of Copy Number Variations and Genetic Variants in POI
Acronym: POI
Status: Recruiting | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Scaruffi, Principal investigator, Ospedale Policlinico San Martino
Other Study IDs: POI genome
Record Dates: First submitted 2022-03-17; First posted 2022-04-14 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Primary Ovarian Insufficiency
Keywords: Premature ovarian failure; array-CGH; NGS
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sporadic POI: Idiopathic, sporadic POI Caucasian cases. The inclusion criteria will be:
  * age at diagnosis <38 years;
  * a normal 46,XX karyotype (no FRM1 premutation);
  * at least one marker of ovarian reserve not age-appropriate:
    * baseline FSH levels > cut-off [1] and/or
    * age-specific AMH < cut-off [2] and/or
    * AFC < 5; and/or
  * cancellation of a PMA cycle because of poor response (<3 follicles) to high-dose gonadotrophins (250 U/die) and/or
  * retrieval of < 4 oocytes in response to high-dose stimulation protocols (3000 U of gonadotrophins).
- Familial POI: Familial POI cases and not-affected members of pedigrees.

SUMMARY:
Primary ovarian insufficiency (POI), also known as premature ovarian failure, is an ovarian defect characterized by the premature (before the age of 40 years) depletion of ovarian follicles. POI affects about 1% of women, reaching 30% in some familial cases.

This heterogeneous disorder is characterized by progressive cessation of the ovarian function with temporary or intermittent amenorrhea associated with elevated serum FSH concentration and low AMH dosage. Low serum AMH dosage is able to detect a diminished ovarian pool occurring before the onset of FSH elevation and the ultimate deficiency leading to amenorrhea.

POI causes infertility and a poor ovarian response in IVF stimulations, and it has important health consequences for affected patients, including psychological distress, infertility, osteoporosis, autoimmune disorders, ischaemic heart disease.

Although the cause of POI remains unknown in about 80% of the cases, several mechanisms have been proposed to explain ovarian dysfunction. Currently, a wide spectrum of causes has been linked to POI, including genetic, autoimmune, infectious, or iatrogenic ones.

Genetic causes are highly heterogeneous and might explain at least some of the sporadic idiopathic cases, which comprise 50-90% of cases. Ten to fifteen percent of cases are X-linked abnormalities, mainly Turner Syndrome (45,X) or X structural abnormalities such as X deletions, X inversions, isochromosomes or X-autosome translocations. Also fragile X mental retardation 1 (FMR1) gene permutation (defined as having 55 to 200 CGG repeats in the 5' untranslated region of the gene) is another frequent genetic etiology.

Irrespectively, the majority of cases remains idiopathic, and identifying precise causative genes for POI has been challenging.

DETAILED DESCRIPTION:
Although in the last decades an increasing number of aberrant genes involved in POI were identified, currently only a minority of affected women can be explained at gene level. Elucidating the biology of the premature declining ovarian function is paramount to develop better testing and treatment strategies for affected women in the future.

Importantly, two clinical features remain unexplained: i) the overall sporadic nature of POI, and ii) observations of patients harboring the identical mutation yet developing POI either early in life (puberty) or later (< 40 years old). Therefore, the investigators postulate that defects affecting more than one gene might explain this variability. Based on investigators' preliminary data and literature reports, it is likely that a synergistic effect of several variant/gene abnormalities may underlie the idiopathic POI phenotype.

The investigators hypothesize that different genome-wide strategies (namely, high resolution array-CGH and WES) may discover genetic variants without the limitation of a single candidate or a panel of candidates, and thus are more promising for explanation of the genetic heterogeneity of POI and elucidating the pathogenic mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* age at diagnosis <38 years;
* a normal 46,XX karyotype (no FRM1 premutation);
* at least one marker of ovarian reserve not age-appropriate:

  * baseline FSH levels > cut-off [1] and/or
  * age-specific AMH < cut-off [2] and/or
  * AFC < 5; and/or
* cancellation of a PMA cycle because of poor response (<3 follicles) to high-dose gonadotrophins (250 U/die) and/or
* retrieval of < 4 oocytes in response to high-dose stimulation protocols (3000 U of gonadotrophins).

Exclusion Criteria:

* patients with POI-related conditions, such as ovarian surgery or previous chemo- or radio-therapy; endometriosis or known autoimmune or metabolic diseases.

Ages: 15 Years to 38 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Idiopathic, sporadic and familial POI cases.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-01-31; Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of putative POI-related genes. | Year 1-20
  Genomic imbalances (<5 Mb in size: copy number variations (CNVs) as micro-deletions and micro-duplications) will be detected in sporadic idiopathic POI patients with the purpose to clarify the role of CNVs in POI pathogenesis and to better unveil both novel candidate genes and pathogenic mechanisms
Identification of genetic variants co-segregated with phenotype. | Year 1-20
  Novel genetic variants not previously anticipated will be found: given the variants co-segregate with phenotype, whole-exome sequencing approach in consanguineous and POI pedigrees will identify the causative gene and variants that cause the phenotype.
To combine array-CGH and WES data mining. | Year 1-20
  The cumulative effect of different genes/variants will be considered in support of the polygenicity of POI and its heterogeneous phenotype (primarily, the sporadic and familial ones).

CONTACTS AND LOCATIONS:
Overall Officials: Paola Scaruffi, Principal Investigator — Ospedale San Martino; Paola Anserini, Study Director — Ospedale San Martino
Locations (1):
- UOS Fisiopatologia della Riuproduzione Umana, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided